CLINICAL TRIAL: NCT05830071
Title: A Randomized, Double-blind, Positive and Placebo-controlled, Single-dose, Crossover Study of the Effects of CHF5993 pMDI (BDP/FF/GB) at the Proposed Therapeutic and Supratherapeutic Doses, on the Cardiovascular Safety in Healthy Subjects
Brief Title: A Thorough QT (TQT) Study of CHF5993 pMDI in Healthy Volunteers (HV)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: CLI-05993AB7-03
Record Dates: First submitted 2023-03-28; First posted 2023-04-26 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — Beclomethasone; Formoterol Fumarate; Glycopyrrolate; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Single therapeutic dose of CHF5993 (BDP/FF/GB) (Experimental): Dose: BDP/FF/GB 100/6/12.5 μg, single dose inhalation via pressurized metered dose inhaler (2 puffs from 1 BDP/FF/GB 100/6/12.5 μg pMDI + 2 puffs from 3 placebo pMDI)
  Interventions: Drug: CHF5993; Drug: CHF5993 Placebo
- Single supra-therapeutic dose of CHF5993 (BDP/FF/GB) (Experimental): Dose: BDP/FF/GB 800/48/100 μg single dose inhalation, via pressurized metered dose inhaler (8 puffs from 4 BDP/FF/GB 100/6/12.5 μg pMDI)
  Interventions: Drug: CHF5993
- Single supra-therapeutic dose CHF5259 (GB) (Experimental): Dose: GB 100 μg single dose inhalation, via pressurized metered dose inhaler (8 puffs from 4 GB 12.5 μg pMDI)
  Interventions: Drug: CHF5259
- Single dose Placebo (Placebo Comparator): Dose: placebo single dose inhalation, via pressurized metered dose inhaler 8 puffs from 4 CHF5993 placebo pMDI
  Interventions: Drug: CHF5993 Placebo
- Moxifloxacin (Active Comparator): Dose: moxifloxacin 400 mg single dose, for oral use - open label treatment (1 tablet of moxifloxacin 400 mg PO)
  Interventions: Drug: Moxifloxacin 400mg

INTERVENTIONS:
Drug: CHF5993 — BDP/FF/GB 100/6/12.5 μg pMDI
  Other Names: beclometasone dipropionate /formoterol fumarate/glycopyrronium bromide; BDP/FF/GB
  Arms: Single supra-therapeutic dose of CHF5993 (BDP/FF/GB); Single therapeutic dose of CHF5993 (BDP/FF/GB)
Drug: CHF5259 — GB 12.5 μg pMDI
  Other Names: glycopyrronium bromide; GB
  Arms: Single supra-therapeutic dose CHF5259 (GB)
Drug: Moxifloxacin 400mg — 400 mg Oral Tablets
  Other Names: Moxifloxacin hydrochloride
  Arms: Moxifloxacin
Drug: CHF5993 Placebo — placebo pMDI
  Other Names: BDP/FF/GB Placebo
  Arms: Single dose Placebo; Single therapeutic dose of CHF5993 (BDP/FF/GB)

SUMMARY:
The purpose of this study is to evaluate the potential for cardiac repolarization, according to electrocardiographic monitoring (including QT and QTc intervals), of two dose levels of CHF5993 pMDI (beclomethasone dipropionate/formoterol fumarate/glycopyrronium bromide (BDP/FF/GB)) and of one dose of CHF5259 (GB) in healthy subjects compared to moxifloxacin and placebo.

DETAILED DESCRIPTION:
The main purpose of this study is to evaluate the effect of a single supratherapeutic dose of inhaled BDP/FF/GB on cardiovascular safety. The secondary purposes of the study are to: 1) evaluate the effect of a single supratherapeutic dose of inhaled BDP/FF/GB and GB on cardiovascular safety; 2) establish assay sensitivity by demonstrating the effect of a single oral dose of 400 mg moxifloxacin on cardiovascular safety; 3) determine the pharmacokinetics (PK) of single, inhaled therapeutic and supratherapeutic BDP/FF/GB doses and supratherapeutic GB dose; 4) determine if there is a relationship between the duration of the QTc intervals and the plasma concentrations of the B17MP (beclomethasone 17monopropionate active metabolite of BDP), FF and GB following the administration of BDP/FF/GB and GB pMDIs; 5) generate additional safety and tolerability information.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject's written informed consent;
* 18-55 years of age;
* Ability to understand the study procedures, the risks involved and ability to be trained to use the inhalers correctly;
* Body Mass Index (BMI) between 18 and 32 kg/m2 extremes inclusive;
* Non- or ex-smokers who smoked < 5 pack years and stopped smoking > 1 year prior to screening;
* Good physical and mental status, determined on the basis of the medical history and a general clinical examination;
* Vital signs within normal limits at screening and prior to randomization: Diastolic BP 40-89 mmHg, Systolic BP 90-139 mmHg extremes included (mean value of three measures). Body temperature < 37.5°C;
* 12 -lead digitized Electrocardiogram (12-lead ECG) in triplicate considered as normal (40 ≤ Heart rate ≤ 110bpm, 120 ms ≤ PR ≤ 220 ms, QRS ≤ 110 ms, QTcF ≤ 450 ms);
* Lung function measurements within normal limits (normal values: forced expiratory volume in the 1st second [FEV1]/forced vital capacity [FVC] > 0.70 and FEV1 > 80% predicted);
* Female subjects of non-child bearing potential or females of child bearing potential with negative pregnancy test; and acceptable contraceptive methods.

Key Exclusion Criteria:

* Participation in another clinical trial where investigational drug was received and last investigations within the last 8 weeks;
* Clinically significant abnormal standard ECG at screening;
* Clinically relevant and uncontrolled respiratory, cardiac, hepatic, gastrointestinal, renal, endocrine, metabolic, neurologic, or psychiatric disorders that may interfere with successful completion of this protocol;
* Subjects with medical diagnosis of narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that in the opinion of the investigator would prevent use of anticholinergic;
* Subjects with history of breathing problems (i.e., history of asthma including childhood asthma);
* Positive urine test for cotinine;
* Intake of non-permitted concomitant medications in the predefined period prior to screening or prior to randomization, or the subject is expected to take non-permitted concomitant medications during the study;
* Presence of any current infection, or previous infection that resolved less than 7 days prior to screening or to randomization;
* Known intolerance and/or hypersensitivity to any of the excipients contained in the formulation used in the trial;
* Women who are pregnant or lactating;
* Use of any kind of smoking electronic devices within 6 months before Screening.

Other inclusion/exclusion criteria as defined by the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Effect of BDP/FF/GB pMDI at therapeutic dose on the heart rate-corrected QT interval based on the Fridericia's correction (QTcF). | time 0 (pre-dose) to 24 hours
  Placebo-adjusted change in QTc interval based on the Fridericia's correction (ΔΔQTcF) after dosing CHF5993 pMDI (200/12/25 μg). Through digitised 12-lead ECG, extracted from 12-Lead Holter ECG.

SECONDARY OUTCOMES:
Effect of BDP/FF/GB pMDI and GB pMDI at supra-therapeutic dose on the heart rate-corrected QT interval based on the Fridericia's correction (QTcF). | time 0 (pre-dose) to 24 hours
  Placebo-adjusted change from baseline in QTc interval based on the Fridericia's correction (ΔΔQTcF) after dosing CHF5993 pMDI (800/48/100 μg) and GB pMDI (100 μg). Through digitised 12-lead ECG, extracted from 12-Lead Holter ECG.
Assay sensitivity by demonstrating the effect of a single oral therapeutic dose of moxifloxacin on QTcF. | time 0 (pre-dose) to 6 hours
  Placebo-adjusted change from baseline in QTc interval based on the Fridericia's correction (ΔΔQTcF) after dosing 400 mg of moxifloxacin. Through digitised 12-lead ECG, extracted from 12-Lead Holter ECG
Effect of BDP/FF/GB pMDI at therapeutic and supra-therapeutic dose and of GB pMDI at supra-therapeutic dose on Hearth Rate (HR). | time 0 (pre-dose) to 24 hours
  Placebo-adjusted change from baseline of HR (ΔΔHR) after dosing BDP/FF/GB pMDI (200/12/25 μg and 800/48/100 μg) and GB pMDI (100 μg) will be summarized by means of descriptive statistics at each analysis time point and by treatment. Through digitised 12-lead ECG, extracted from 12-Lead Holter ECG.
Effect of BDP/FF/GB pMDI at therapeutic and supra-therapeutic dose and of GB pMDI at supra-therapeutic dose on PR interval (PR). | time 0 (pre-dose) to 24 hours
  Placebo-adjusted change from baseline of PR (ΔΔPR) after dosing BDP/FF/GB pMDI (200/12/25 μg and 800/48/100 μg) and GB pMDI (100 μg) will be summarized by means of descriptive statistics at each analysis time point and by treatment. Through digitised 12-lead ECG, extracted from 12-Lead Holter ECG.
Effect of BDP/FF/GB pMDI at therapeutic and supra-therapeutic dose and of GB pMDI at supra-therapeutic dose on QRS interval (QRS). | time 0 (pre-dose) to 24 hours
  Placebo-adjusted change from baseline of QRS (ΔΔQRS) after dosing BDP/FF/GB pMDI (200/12/25 μg and 800/48/100 μg) and GB pMDI (100 μg) will be summarized by means of descriptive statistics at each analysis time point and by treatment. Through digitised 12-lead ECG, extracted from 12-Lead Holter ECG.
Effect of BDP/FF/GB pMDI at therapeutic and supra-therapeutic dose and of GB pMDI at supra-therapeutic dose on individual-corrected QT interval (QTcI) | time 0 (pre-dose) to 24 hours
  Placebo-adjusted change from baseline in individual-corrected QT interval (ΔΔQTcI) after dosing BDP/FF/GB pMDI (200/12/25 μg and 800/48/100 μg) and GB pMDI (100 μg). Through digitised 12-lead ECG, extracted from 12-Lead Holter ECG.
Effect of moxifloxacin at therapeutic dose on individual-corrected QT interval. | time 0 (pre-dose) to 6 hours
  Placebo-adjusted change from baseline in individual-corrected QT interval (ΔΔQTcI) after dosing 400 mg of moxifloxacin. Through digitised 12-lead ECG, extracted from 12-Lead Holter ECG.
Changes in T-wave morphology and U-wave presence. | time 0 (pre-dose) to 24 hours
  Frequency of treatment-emergent changes in T-wave morphology and U-wave presence after dosing BDP/FF/GB pMDI (200/12/25 μg and 800/48/100 μg) and GB pMDI (100 μg). Through digitised 12-lead ECG, extracted from 12-Lead Holter ECG.
Analysis of categorical outliers of Hearth Rate (HR), PR interval (PR), QRS interval (QRS) and QTcF interval (QTcF), after BDP/FF/GB pMDI dosing at therapeutic and supra-therapeutic dose, and after GB dosing at supra-therapeutic dose. | time 0 (pre-dose) to 24 hours
  Results of categorical outliers will be summarized by treatment in frequency tables reporting: counts and percentages for number of subjects and number of time points with 1) abnormal actual QTcF values, and 2) abnormal change from baseline of HR, PR, QRS and QTcF. Through digitised 12-lead ECG, extracted from 12-Lead Holter ECG.
Analysis of Maximum plasma concentration (Cmax), pharmacokinetic parameter of FF, GB, BDP and B17MP | time 0 (pre-dose) to 24 hours
  Analysis of Cmax after dosing BDP/FF/GB pMDI (200/12/25 μg and 800/48/100 μg) and GB pMDI (100 μg).
Analysis of Area under the curve from 0 to 12 hours post-dose (AUC0-12), pharmacokinetic parameter of FF, GB, BDP and B17MP | time 0 (pre-dose) to 24 hours
  Analysis of AUC0-12, after dosing BDP/FF/GB pMDI (200/12/25 μg and 800/48/100 μg) and GB pMDI (100 μg).
Analysis of Area under the plasma concentration-time curve from time 0 to time t (AUC0 t), pharmacokinetic parameter of FF, GB, BDP and B17MP | time 0 (pre-dose) to 24 hours
  Analysis of AUC0-t after dosing BDP/FF/GB pMDI (200/12/25 μg and 800/48/100 μg) and GB pMDI (100 μg).
Analysis of Area under the curve from time 0 to infinity (AUC0-∞), pharmacokinetic parameter of FF, GB, BDP and B17MP | time 0 (pre-dose) to 24 hours
  Analysis of AUC0-∞ after dosing BDP/FF/GB pMDI (200/12/25 μg and 800/48/100 μg) and GB pMDI (100 μg).
Analysis of Time to maximum plasma concentration (tmax), pharmacokinetic parameter of FF, GB, BDP and B17MP | time 0 (pre-dose) to 24 hours
  Analysis of tmax, after dosing BDP/FF/GB pMDI (200/12/25 μg and 800/48/100 μg) and GB pMDI (100 μg).
Analysis of Terminal half-life (t1/2), pharmacokinetic parameter of FF, GB, BDP and B17MP | time 0 (pre-dose) to 24 hours
  Analysis of t1/2, after dosing BDP/FF/GB pMDI (200/12/25 μg and 800/48/100 μg) and GB pMDI (100 μg).
Incidence of Adverse events | from study start through study completion, an average of 4 months
  Number and percentage of subjects with at least one event and number of treatment emergent events
Incidence of Adverse Drug Reactions | from study start through study completion, an average of 4 months
  Number and percentage of subjects with at least one event and number of treatment emergent events
Change of systolic and diastolic blood pressure | from study start through study completion, an average of 4 months
  Number and percentage of subjects with with abnormal changes from baseline
Body temperature abnormal values | from study start through study completion, an average of 4 months
  Number and percentage of subjects with at least one event and number of treatment emergent events
Abnormal results of physical examinations | from study start through study completion, an average of 4 months
  Number and percentage of subjects with at least one event and number of treatment emergent events
Abnormal clinical chemistry and haematology laboratory tests | from study start through study completion, an average of 4 months
  Number and percentage of subjects with at least one event and number of treatment emergent events

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, MDCM/M.SC(A), Principal Investigator — PAREXEL Baltimore Early Phase Clinical Unit
Locations (1):
- PAREXEL Baltimore Early Phase Clinical Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No